CLINICAL TRIAL: NCT05899348
Title: iTEST: Introspective Accuracy as a Novel Target for Functioning in Psychotic Disorders
Acronym: iTEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The University of Texas at Dallas (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Colin Depp, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R61MH129379-01A1 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- iTEST (Experimental)
  Interventions: Behavioral: iTEST

INTERVENTIONS:
Behavioral: iTEST — iTEST is a computerized training intervention delivered on a mobile device that is coupled with individual contacts with a therapist/coach. The mobile components train in improving participant's ability to form accurate judgments about their performance and their rate of functional activities. The intervention involves coaching coupled with automated training that is delivered on a mobile device. The automated training involves daily cognitive tests in which the goal for treatment is to improve judgments of accuracy of self-assessment, and coaching is aimed at applying improving metacognitive awareness to every day activities.

SUMMARY:
People with psychotic disorders experience a high level of functional disability, and a major contributor to this disability is introspective accuracy, which is defined as inaccurate judgements of one's abilities and performance on tasks. Yet, no intervention has directly targeted introspective accuracy for psychotic illnesses. This trial will evaluate a new intervention, called iTEST, that uses mobile devices to train people with psychotic disorders to improve introspective accuracy and, ultimately, functional outcomes

DETAILED DESCRIPTION:
This NIH-supported clinical trial is the first phase of a two phase program, funded by Development of Psychosocial Therapeutic and Preventive Interventions for Mental Disorders, R61/R33. The overarching goal is to evaluate a new blended mobile intervention that is aimed at improving introspective accuracy (IA) in people with psychotic disorders, with the ultimate goal of improving functional outcome. Introspective accuracy is the degree to which one's self-assessment of performance or abilities corresponds with objective data. Recent research indicates that poor IA is an independent predictor of functional disability. Yet, there are currently no treatments that directly target IA. Basic experimental research and other lines of evidence suggest IA is malleable, and that improvement in task-based IA transfers to untrained tasks. This project's premise is that task-based IA training could be delivered in a remote mobile health format and coupled with coaching in applying improved IA to real-world functional behaviors, creating a novel avenue for functional rehabilitation in psychotic disorders. The investigators have developed and completed usability testing of iTEST, a novel blended IA targeted mobile intervention. iTEST integrates graduated drill-and-practice training in IA delivered on a mobile device with personalized coaching in applying IA to everyday compensatory behaviors. In the R61 phase trial here, the investigators will recruit people with psychotic disorders with at least minimal functional impairment. The investigators will conduct an open trial of iTEST, evaluating whether the intervention leads to clinically significant changes in task-based IA along with transfer to an untrained task (target mechanisms). The investigators will also determine the dose of intervention needed to achieve clinically significant improvement in IA targets, by evaluating change at 8, 12, or 16 weeks. The go/no go criteria for this trial are 75% adherence and clinically significant increases in introspective accuracy. A total of 60 persons who are diagnosed with schizophrenia or schizoaffective disorder will be recruited into this trial

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary informed consent to participate and capacity to consent as measured by the UCSD Brief Assessment of Capacity to Consent (UBACC)
2. Age 18 to 65;
3. DSM-5 diagnosis of schizophrenia or schizoaffective disorder based on a structured diagnostic interview and available medical record review;
4. ≥ 6th grade reading level on the Wide Range Achievement Test-4 Reading subtest (needed to read instructions on device);
5. Stable co-treatments (no hospitalizations or medication class changes in 2 months before enrollment). The investigators will determine symptom and medication stability by best-estimate history with information from medical records;
6. Availability of a clinician (staff member, case manager, other mental health clinician) or close associate (family member, friend) with at least monthly contact who can be their informant
7. Minimum level of functional impairment based on milestones, excluding participants who are full-time employed and financially responsible for their household.

Exclusion Criteria:

1. Greater than moderate disorganization on the Positive and Negative Syndrome Scale (P2-Disorganization item >5)
2. DSM-5 alcohol or substance dependence in past 3 months based on interview
3. Level of care required interferes with outpatient therapy (e.g., hospitalized; severe medical illness); 4) Unable to adequately see or manually manipulate a smartphone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Trained Introspective Accuracy | Change from Baseline to 16 week follow up assessment
  Introspective accuracy is measured daily basis from baseline to 16 weeks (average of introspective accuracy determined from self-reported estimated correct on the Variable Length List Learning Memory Test; Mobile Electronic Test of Emotion Recognition and actual correct). Each day, participants complete tasks in which the can obtain a number of correct responses in guessing the emotion depicted on a picture of a human face and remembering a list of words provided to them. Participants are then asked to guess how many items correctly identified and introspective accuracy is the absolute value of the difference between the guessed correct and actual correct. This number can range from zero to ten and lower scores reflect better introspective accuracy. There are two measures of introspective accuracy (one from a facial recognition task and the other from a word list task) and these are averaged within each day.
Untrained Introspective Accuracy on WCST | Change from Baseline to 16 week follow up assessment
  The Metacognitive Wisconsin Card Sorting Test (WCST) is a secondary measure of introspective accuracy and involves the completion of the standard neuropsychological task (WCST) with simultaneous questions about the participants judgment of correctness. The primary unit of analysis is the difference between self-assessed correct and actual correct responses.
Adherence | Change over 16 weeks
  Completion of daily mobile prompts divided by the number possible

SECONDARY OUTCOMES:
Specific Level of Function Scale (Informant Version) | Change from Baseline Assessment to 16 week follow up Assessment
  The Specific Level of Functioning (SLOF) is an informant rated scale of functioning in the community. The measure includes 43 items that address current work, self-care, social and related functional capacities. The summary variable is the higher order functional factor which combines work, independent living, and social functional capacity. The maximum score is 215 and the minimum score is 43, with higher scores reflective of better functioning

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - University of Texas at Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
A condition of funding is that IPD is made available to other researchers through the National Data Archive of the NIMH. The investigative team will deposit and share data in the NIMH National Data Archive and the investigative team has budgeted staff time of 100 hours per year to accomplish the preparation, curation, and uploading of semiannual de-identified data as the study progresses (linked with Global Unique Identifiers) to the online system in collaboration with NIH staff. • The investigative team will develop documents and tools to support this dissemination, in particular for the sharing ecological momentary assessment data which presents data management challenges in its volume and complexity, including within-person aggregation scripts that can be used to analyze the data at the day and week level. IPD that will be shared include all de-identified study data
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available by September 2025, which is within 6 months of the conclusion of the award. This is consistent with NIMH policy on the timing of data sharing and data will be shared in perpetuity.
Access Criteria: Individuals seeking data access it through the National Data Archive wherein access controlled by the NIH

REFERENCES:
- [Derived] Berretta SA, Abaya N, Parrish E, McBride LE, Moore RC, Ackerman R, Harvey PD, Pinkham AE, Depp CA. Protocol for evaluation of iTEST, a novel blended intervention to enhance introspective accuracy in psychotic disorders. NPP Digit Psychiatry Neurosci. 2025;3(1):5. doi: 10.1038/s44277-024-00024-7. Epub 2025 Feb 14. PMID 39959603